CLINICAL TRIAL: NCT05876013
Title: Reduced Knee Flexion Strength 18 Years After ACL Reconstruction in Hamstring Group
Brief Title: Reduced Knee Flexion Strength 18 Years After ACL Reconstruction in Hamstring Group Compared to Patellar Tendon Group
Acronym: Studie ACL
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other); Haraldsplass Deaconess Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 391796
Record Dates: First submitted 2023-04-17; First posted 2023-05-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: ACL; ACL Injury; Cruciate Ligament Rupture; ACL Tear; Surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BPTB group: Bone-patellar tendon- bone graft used for ACL reconstruction.
  Interventions: Procedure: ACL reconstruction
- Hamstring group: Double-looped semitendinosus and gracilis graft used for ACL reconstruction
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — Randomized between hamstring and patellar tendon graft
  Other Names: Graft choice,

SUMMARY:
Background: Bone-patellar tendon-bone (BPTB) and a double-looped semitendinosus gracilis (hamstring group) graft are commonly used for ACL reconstruction. Short-term and mid-term studies show little to no significant difference between the two groups, and there are a few long term studies to compare results between the two grafts.

Purpose: To compare the results after using either BPTB grafts or hamstring grafts 18 years after ACL reconstruction.

Study design: Randomized controlled trial; Level of evidence II. Methods: 114 patients with ACL rupture between 2001 and 2004 were randomized to reconstruction with either BPTB graft or a hamstring graft. Patients were operated at four major hospitals. The 18-year follow-up evaluation included isokinetic testing of muscle strength, patient-reported outcome measures, clinical knee examination and an assessment of radiological osteoarthritis using the Kellgren-Lawrence classification.

Hypothesis:Hypothesis is that there will be no difference in the long-term outcome between the two groups, as well hypothesis of no difference in patients with prosthesis after ACL reconstruction, arthrosis difference in operated knees and the rate of graft failure between the two groups. Previous follow-up studies showed a significant difference in total flexion work between the two groups, so detecting a persistent difference between the groups will be point of interest.

DETAILED DESCRIPTION:
Introduction Rupture of the anterior cruciate ligament (ACL) is a common soft-tissue knee injury, and has increased in number over the last twenty years. Reconstructing the ligament may be important for maintaining the stability and preventing further damaging of the knee. The two most commonly used grafts in reconstructions are the autologous patellar tendon grafts and hamstring tendon grafts There is yet to be a universally established agreement regarding which reconstruction method of an ACL is preferred. The method using the central third of the patellar tendon with proximal and distal bone blocks as the replacement has been used since the late 80s and is well documented with good results. When the technique using the hamstring tendon grafts was introduced, its popularity increased. Arguments favoring each of the methods depend on which variables one values the most. In some studies, the patellar tendon group reported problems regarding anterior knee pain and decreased sensitivity of the knee, whereas for the hamstring tendon group there was reported increased weakness of the hamstring muscles and knee laxity. However, the overall assessment and satisfaction in multiple short-term/semi-long studies have shown little to no difference .

The aim of this prospective randomized multicenter study is to compare the use of bone-patellar tendon-bone (BPTB) grafts and double-looped semitendinosus gracilis (DLSG) grafts for reconstruction of the anterior cruciate ligament, 17-20 years after the surgery. The null hypothesis is that there will be no significant differences at this long-term follow-up evaluation between the two methods.

Method and material of the first study- Drogset et al. recruited 115 patients with rupture of the anterior cruciate ligament in the period of 2001-2004, and randomized them to either reconstruction with bone-patellar tendon-bone (BPTB) grafts fixed with metal interference screw graft, or double-looped semitendinosus gracilis (DLSG) grafts fixed with Bone Mulch Screws and WasherLoc Screws. The surgeries were performed at four different hospitals.

After one and two years, the patients were examined by an independent observer, using a series of objective tests, as well as recording the patients' subjective opinion of their knee function. The subjective tests used were Tegner's activity score, Lysholm's functional score and Modified Cincinnati Score. The objective tests used were Lachmann's test, pivot shift and KT-1000, as well as Cybex and Biodex to measure muscle strength.

Method and material- The present study is a long-term follow-up of a prospective randomized multicenter study. The patient recorded outcome scores will be Tegner's activity score, Lysholms's functional score and the Knee injury Osteoarthritis Outcome Score (KOOS). The examinations include Lachmann's test, pivot shift and KT-1000. We also plan to include radiographs to evaluate the degree of arthrosis 17-20 years after the surgery, and Cybex or Biodex to examine the hamstring and quadriceps strength. The radiographic positioning will be knee AP weight-bearing standing bilateral and lateral view, as well as skyline projection. The Kellgren-Lawrence classification will be used to assess the degree of osteoarthritis.

Even though 115 patients were included in the original study, we will only attempt to contact 114 due to lost inclusion-papers between the 2-year and 7-year follow-up [8]. During the spring of 2022, the patients will receive an invite to participate in the follow-up study. Following this, patients will be contacted to uncover different circumstances that might exclude certain patients from the clinical assessment. This includes revision of the reconstruction in question, total knee replacement or total knee arthroplasty, and if the knee had been injured beforehand. The clinical examination will be carried out by both a medical student and an experienced orthopedic surgeon. Hopefully all the patients will be examined over the course of two days at each location, and if needed, the rest will be examined at a later date.

Hypothesis- Current hypothesis is that there will be no difference in the long-term outcome between the two groups. However, it will be interesting to see how many patients have received a prosthesis, and how many patients struggle with arthrosis. As the previous follow-up studies showed a significant difference in total flexion work between the two groups, we will be interested in detecting a persistent difference between the groups.

Another interesting aspect will be the rate of graft failure between the two groups.

Feasibility- The strength of the study is the randomization and the long follow-up period of 17-20 years. The possible limitations are the fact that there may be a problem recruiting enough patients to the follow-up, and that it might not be able to get x-rays of the patients at the different hospitals, as this is a matter of cost and availability. In addition, the different hospitals may not have a Biodex available.

Publicity plan- The goal for the paper is to be published in an international journal and probably be presented at conferences. For article, that hopefully will be published in journals, Marko Popovic will stand as first author, and Julie Holen and Julie Myhre as contributing authors. Jon Olav Drogset will be listed last, as the main supervisor.

Ethics- The REK-application was submitted on the 24th of December 2021. Application number: 391796. Additionally, the project will be reported to NSD when the REK-application is approved.

ELIGIBILITY:
Inclusion Criteria:

* Primary reconstructions of isolated ACL-ruptures. Surgery at least 6 weeks after injury. Age 18-45 years.
* The patient must understand and accept the written consent. The written consent must be signed by the patient before surgery.
* Normal two-plane X-ray of the knee.

Exclusion Criteria:

->5mm + chronic MCL-injury in the same knee.

* Patient with major additional injury in the knee: combined instability, cartilage injuries Outerbridge grade 3-4 and at least 1cm in diameter on the femoral condyle and major meniscal lesions with meniscal repairs.
* Patients having problems following the protocol.
* The patient does not understand the written consent or will not sign it.
* Patients with a history of alcohol or drug abuse the last three years.
* The patient has received any investigational drugs within 30 days prior to admittance to this study.
* The patient has O.A., podagra, RA, Bechterew's disease or chondrocalcinosis.
* The patient has malalignment with more than 5 degrees valgus and no varus compared to a normal knee.
* The patient has patellofemoral instability.
* The patient is obese with BMI>30.
* The patient has a present or former serious illness that makes follow-up or rehabilitation of the patient difficult.
* Former major surgical procedures in the same knee, including prosthesis.
* Treated or untreated anterior cruciate ligament injury in the other knee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Norwegian citizens. Patients from Trondelag county operated in Trondheim (StOlav Hospital), patients from Oslo operated at Lovisenberg Diaconal Hospital Oslo, patients from Hordaland operated at Haraldsplass Deaconess Hospital Bergen. Few patients from other counties who wanted operation at spesific hospital were also included if inclusion criteria were met.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
KT-1000 arthrometer | Examination day, 1 day.
  KT-1000 test- The KT1000 arthrometer was designed to measure the anterior translation of the tibia while maintaing the femur in position. The results obtained provide an objective diagnostic of the state of the ACL to the medical practitioner.

SECONDARY OUTCOMES:
Gonarthrosis measurement | Examination day, 1 day
  Kellgren Lawrence classification was used to determine grade of gonarthrosis in operated and non-operated knee, both in patello-femoral and tibio-femoral joint.
Biodex isokinetic testing | Examination day, 1 day.
  Biodex is a isokinetic machine used to measure muscle strength and identify weaknesses in certain muscle groups. It can be used in different degrees to measure muscle strength in different positions of the joint.
KOOS score | Examination day, 1 day
  The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems. This direction, 100 indicating no problems, is common in orthopaedic instruments and generic measures like the SF-36.
Lysholm's functional score | Examination day, 1 day
  In the modified Lysholm system the maximum score is 100 points, in which: 91 to 100 points is considered excellent; 84 to 90, good; 65 to 83, fair; and 64 or less, unsatisfactory. Lysholm's system is an evaluation system that includes three functional criteria and five subjective criteria.
Tegner's activity score | Examination day, 1 day.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Pivot shift test | Examination day, 1 day.
  Pivot shift test- positive test is indicated by subluxation of the tibia while the femur rotates externally followed by a reduction of the tibia at 30-40 degrees of flexion.
Lachmann test | Examination day, 1 day.
  Lachmann test- Anterior translation of the tibia associated with a soft or a mushy end-feel indicates a positive test. More than about 2mm of anterior translation compared to the uninvolved knee suggests a torn ACL ("soft end-feel"), as does 10mm of total anterior translation.

CONTACTS AND LOCATIONS:
Overall Officials: Jon O. Drogset, PhD, Study Chair — St Olav Hospital Trondheim
Locations (1):
- St Olav Hospital, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourke HE, Salmon LJ, Waller A, Patterson V, Pinczewski LA. Survival of the anterior cruciate ligament graft and the contralateral ACL at a minimum of 15 years. Am J Sports Med. 2012 Sep;40(9):1985-92. doi: 10.1177/0363546512454414. Epub 2012 Aug 6. PMID 22869626
- [Background] Leys T, Salmon L, Waller A, Linklater J, Pinczewski L. Clinical results and risk factors for reinjury 15 years after anterior cruciate ligament reconstruction: a prospective study of hamstring and patellar tendon grafts. Am J Sports Med. 2012 Mar;40(3):595-605. doi: 10.1177/0363546511430375. Epub 2011 Dec 19. PMID 22184280
- [Background] Freedman KB, D'Amato MJ, Nedeff DD, Kaz A, Bach BR Jr. Arthroscopic anterior cruciate ligament reconstruction: a metaanalysis comparing patellar tendon and hamstring tendon autografts. Am J Sports Med. 2003 Jan-Feb;31(1):2-11. doi: 10.1177/03635465030310011501. PMID 12531750
- [Background] Gifstad T, Foss OA, Engebretsen L, Lind M, Forssblad M, Albrektsen G, Drogset JO. Lower risk of revision with patellar tendon autografts compared with hamstring autografts: a registry study based on 45,998 primary ACL reconstructions in Scandinavia. Am J Sports Med. 2014 Oct;42(10):2319-28. doi: 10.1177/0363546514548164. Epub 2014 Sep 8. PMID 25201444
- [Background] Gifstad T, Sole A, Strand T, Uppheim G, Grontvedt T, Drogset JO. Long-term follow-up of patellar tendon grafts or hamstring tendon grafts in endoscopic ACL reconstructions. Knee Surg Sports Traumatol Arthrosc. 2013 Mar;21(3):576-83. doi: 10.1007/s00167-012-1947-0. Epub 2012 Mar 10. PMID 22407182
- [Background] Drogset JO, Strand T, Uppheim G, Odegard B, Boe A, Grontvedt T. Autologous patellar tendon and quadrupled hamstring grafts in anterior cruciate ligament reconstruction: a prospective randomized multicenter review of different fixation methods. Knee Surg Sports Traumatol Arthrosc. 2010 Aug;18(8):1085-93. doi: 10.1007/s00167-009-0996-5. Epub 2009 Dec 3. PMID 19956928
- [Background] Herzog MM, Marshall SW, Lund JL, Pate V, Mack CD, Spang JT. Trends in Incidence of ACL Reconstruction and Concomitant Procedures Among Commercially Insured Individuals in the United States, 2002-2014. Sports Health. 2018 Nov/Dec;10(6):523-531. doi: 10.1177/1941738118803616. PMID 30355175
- [Background] Costa-Paz M, Garcia-Mansilla I, Marciano S, Ayerza MA, Muscolo DL. Knee-related quality of life, functional results and osteoarthritis at a minimum of 20 years' follow-up after anterior cruciate ligament reconstruction. Knee. 2019 Jun;26(3):666-672. doi: 10.1016/j.knee.2019.04.010. Epub 2019 May 15. PMID 31103415
- [Background] Risberg MA, Oiestad BE, Gunderson R, Aune AK, Engebretsen L, Culvenor A, Holm I. Changes in Knee Osteoarthritis, Symptoms, and Function After Anterior Cruciate Ligament Reconstruction: A 20-Year Prospective Follow-up Study. Am J Sports Med. 2016 May;44(5):1215-24. doi: 10.1177/0363546515626539. Epub 2016 Feb 24. PMID 26912282
- [Background] Mohtadi NG, Chan DS, Dainty KN, Whelan DB. Patellar tendon versus hamstring tendon autograft for anterior cruciate ligament rupture in adults. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD005960. doi: 10.1002/14651858.CD005960.pub2. PMID 21901700
- [Background] Persson A, Fjeldsgaard K, Gjertsen JE, Kjellsen AB, Engebretsen L, Hole RM, Fevang JM. Increased risk of revision with hamstring tendon grafts compared with patellar tendon grafts after anterior cruciate ligament reconstruction: a study of 12,643 patients from the Norwegian Cruciate Ligament Registry, 2004-2012. Am J Sports Med. 2014 Feb;42(2):285-91. doi: 10.1177/0363546513511419. Epub 2013 Dec 9. PMID 24322979
- [Background] Goldblatt JP, Fitzsimmons SE, Balk E, Richmond JC. Reconstruction of the anterior cruciate ligament: meta-analysis of patellar tendon versus hamstring tendon autograft. Arthroscopy. 2005 Jul;21(7):791-803. doi: 10.1016/j.arthro.2005.04.107. PMID 16012491
- [Background] Holm I, Oiestad BE, Risberg MA, Aune AK. No difference in knee function or prevalence of osteoarthritis after reconstruction of the anterior cruciate ligament with 4-strand hamstring autograft versus patellar tendon-bone autograft: a randomized study with 10-year follow-up. Am J Sports Med. 2010 Mar;38(3):448-54. doi: 10.1177/0363546509350301. Epub 2010 Jan 23. PMID 20097928
- [Background] Mascarenhas R, Tranovich MJ, Kropf EJ, Fu FH, Harner CD. Bone-patellar tendon-bone autograft versus hamstring autograft anterior cruciate ligament reconstruction in the young athlete: a retrospective matched analysis with 2-10 year follow-up. Knee Surg Sports Traumatol Arthrosc. 2012 Aug;20(8):1520-7. doi: 10.1007/s00167-011-1735-2. Epub 2011 Nov 3. PMID 22048746
- [Background] Sajovic M, Vengust V, Komadina R, Tavcar R, Skaza K. A prospective, randomized comparison of semitendinosus and gracilis tendon versus patellar tendon autografts for anterior cruciate ligament reconstruction: five-year follow-up. Am J Sports Med. 2006 Dec;34(12):1933-40. doi: 10.1177/0363546506290726. Epub 2006 Aug 21. PMID 16923826
- [Background] Xie X, Liu X, Chen Z, Yu Y, Peng S, Li Q. A meta-analysis of bone-patellar tendon-bone autograft versus four-strand hamstring tendon autograft for anterior cruciate ligament reconstruction. Knee. 2015 Mar;22(2):100-10. doi: 10.1016/j.knee.2014.11.014. Epub 2014 Dec 11. PMID 25547048
- [Background] Bjornsson H, Samuelsson K, Sundemo D, Desai N, Sernert N, Rostgard-Christensen L, Karlsson J, Kartus J. A Randomized Controlled Trial With Mean 16-Year Follow-up Comparing Hamstring and Patellar Tendon Autografts in Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2016 Sep;44(9):2304-13. doi: 10.1177/0363546516646378. Epub 2016 May 26. PMID 27229354
- [Background] Coffey R, Bordoni B. Lachman Test. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554415/ PMID 32119302
- [Background] Sajovic M, Stropnik D, Skaza K. Long-term Comparison of Semitendinosus and Gracilis Tendon Versus Patellar Tendon Autografts for Anterior Cruciate Ligament Reconstruction: A 17-Year Follow-up of a Randomized Controlled Trial. Am J Sports Med. 2018 Jul;46(8):1800-1808. doi: 10.1177/0363546518768768. Epub 2018 May 9. PMID 29741911
- [Background] Vaudreuil NJ, Rothrauff BB, de Sa D, Musahl V. The Pivot Shift: Current Experimental Methodology and Clinical Utility for Anterior Cruciate Ligament Rupture and Associated Injury. Curr Rev Musculoskelet Med. 2019 Mar;12(1):41-49. doi: 10.1007/s12178-019-09529-7. PMID 30706283
- [Background] Arneja S, Leith J. Review article: Validity of the KT-1000 knee ligament arthrometer. J Orthop Surg (Hong Kong). 2009 Apr;17(1):77-9. doi: 10.1177/230949900901700117. PMID 19398799
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Pinczewski LA, Lyman J, Salmon LJ, Russell VJ, Roe J, Linklater J. A 10-year comparison of anterior cruciate ligament reconstructions with hamstring tendon and patellar tendon autograft: a controlled, prospective trial. Am J Sports Med. 2007 Apr;35(4):564-74. doi: 10.1177/0363546506296042. Epub 2007 Jan 29. PMID 17261567
- [Background] Thompson SM, Salmon LJ, Waller A, Linklater J, Roe JP, Pinczewski LA. Twenty-Year Outcome of a Longitudinal Prospective Evaluation of Isolated Endoscopic Anterior Cruciate Ligament Reconstruction With Patellar Tendon or Hamstring Autograft. Am J Sports Med. 2016 Dec;44(12):3083-3094. doi: 10.1177/0363546516658041. Epub 2016 Aug 4. PMID 27492972
- [Background] Konrads C, Reppenhagen S, Plumhoff P, Hoberg M, Rudert M, Barthel T. No significant difference in clinical outcome and knee stability between patellar tendon and semitendinosus tendon in anterior cruciate ligament reconstruction. Arch Orthop Trauma Surg. 2016 Apr;136(4):521-5. doi: 10.1007/s00402-015-2386-4. Epub 2016 Jan 2. PMID 26725050
- [Background] Bourke HE, Gordon DJ, Salmon LJ, Waller A, Linklater J, Pinczewski LA. The outcome at 15 years of endoscopic anterior cruciate ligament reconstruction using hamstring tendon autograft for 'isolated' anterior cruciate ligament rupture. J Bone Joint Surg Br. 2012 May;94(5):630-7. doi: 10.1302/0301-620X.94B5.28675. PMID 22529082
- [Background] Webster KE, Feller JA, Hartnett N, Leigh WB, Richmond AK. Comparison of Patellar Tendon and Hamstring Tendon Anterior Cruciate Ligament Reconstruction: A 15-Year Follow-up of a Randomized Controlled Trial. Am J Sports Med. 2016 Jan;44(1):83-90. doi: 10.1177/0363546515611886. Epub 2015 Nov 17. PMID 26578718
- [Background] Samuelsen BT, Webster KE, Johnson NR, Hewett TE, Krych AJ. Hamstring Autograft versus Patellar Tendon Autograft for ACL Reconstruction: Is There a Difference in Graft Failure Rate? A Meta-analysis of 47,613 Patients. Clin Orthop Relat Res. 2017 Oct;475(10):2459-2468. doi: 10.1007/s11999-017-5278-9. PMID 28205075
- [Derived] Popovic M, Myhre JR, Holen JIH, Gifstad T, Strand IL, Strand T, Mo IF, Fischer-Bredenbeck C, Drogset JO. Reduced Knee Flexion Strength 18 Years After ACL Reconstruction With Hamstring Tendon Versus Patellar Tendon. Am J Sports Med. 2024 Sep;52(11):2750-2757. doi: 10.1177/03635465241271524. Epub 2024 Sep 2. PMID 39221503

DOCUMENTS (1):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT05876013/Prot_000.pdf